CLINICAL TRIAL: NCT05378412
Title: Efecto Del Modelo "Conmigo, Contigo y Con Todos" (3Cs) en Niños, Niñas y Adolescentes y Sus Profesores en Vaupés, Boyacá y Amazonas
Brief Title: Effect of the 3C Model in Students and Teachers From Vaupés, Boyacá and Amazonas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Saldarriaga Concha (Other)
Collaborators: Pontificia Universidad Javeriana (Other); Ministerio de Ciencia, Tecnología e Innovación (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10085; SIGP 92409 (Other: Ministerio de Ciencias, Tecnología e Innovación)
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Resilience, Compassion

STUDY DESIGN:
Intervention Model Description: This study is based on a mixed-methods experimental design and concurrent triangulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3Cs (Experimental)
  Interventions: Behavioral: 3Cs
- Control (No Intervention)

INTERVENTIONS:
Behavioral: 3Cs — The 3Cs program is an educational strategy aimed at fostering resilience and compassion in people. It is based on improving the mental well-being of the participants by transforming their attitudes and behaviors through increased consciousness.
  Arms: 3Cs

SUMMARY:
This study will evaluate the effectiveness of the "3Cs - Conmigo, Contigo y Con todo" strategy in strengthening resilience and compassion in students and teachers from three regions from Colombia: Vaupés, Amazonas and Boyacá. It will also evaluate its relevance in the design of programs aimed at mental health in educational settings.

DETAILED DESCRIPTION:
Colombia has experienced a long-lasting internal armed conflict that has impacted society at all levels and on people of all ages. This has led to changes in behavior and the way people cope with psychosocial distress. Focusing on children and adolescents, this study aims to assess the effectiveness of the "3Cs - Conmigo, Contigo y Con todo" strategy in strengthening resilience and compassion. The changes in the scores of the CD-RISC and ECOM instruments will be evaluated through a mixed methods analysis that will evaluate the pre and post intervention results and the perception of all the actors involved in the development and implementation of the 3Cs program.

ELIGIBILITY:
Inclusion Criteria:

* Students and teachers from public institutions

Exclusion Criteria:

-

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6000 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
CD-RISC | 36 months
  CD-RISC score
ECOM | 36 months
  ECOM score

IPD SHARING:
Plan to Share IPD: No